CLINICAL TRIAL: NCT02307461
Title: A Phase 1, Open-label, 2-Part Study to Evaluate the Bioequivalence of the Duvelisib Marker-Image Formulation to the Duvelisib Clinical-Trial Formulation and to Assess the Effect of Food on the Pharmacokinetics of IP Duvelisib in Healthy Adult Subjects
Brief Title: Bioequivalence of Duvelisib and Food Effect on Pharmacokinetics of IPI-145
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IPI-145-15
Record Dates: First submitted 2014-11-18; First posted 2014-12-04 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Healthy
Keywords: Phase 1; Bioequivalence; Pharmacokinetics; Food; Healthy Adult
MeSH Terms: interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 Cohort 1 (Experimental): IPI-145 test formulation (capsule) high single dose and IPI-145 reference formulation (capsule) high single dose
  Interventions: Drug: IPI-145 (duvelisib)
- Part 1 Cohort 2 (Experimental): IPI-145 test formulation (capsule) low single dose and IPI-145 reference formulation (capsule) low single dose
  Interventions: Drug: IPI-145
- Part 2 Cohort 3 (Experimental): IPI-145 test formulation (capsule) high single dose administered under fasted and fed conditions
  Interventions: Drug: IPI-145

INTERVENTIONS:
Drug: IPI-145 (duvelisib) — High single oral dose capsule IPI-145 test formulation and IPI-145 reference formulation (capsule) high single oral dose
  Arms: Part 1 Cohort 1
Drug: IPI-145 — Low single oral dose capsule IPI-145 test formulation and IPI-145 reference formulation (capsule) low single oral dose
  Arms: Part 1 Cohort 2
Drug: IPI-145 — High single oral dose IPI-145 test formulation (capsule) with a high-fat meal and without food
  Arms: Part 2 Cohort 3

SUMMARY:
To Evaluate the Bioequivalence of the two formulations of IPI-145 and the Effect of Food on the Pharmacokinetics of IPI-145

DETAILED DESCRIPTION:
This Phase 1, randomized, open-label study of IPI-145 will be conducted in 2 parts.

Part 1 will be conducted in 2 cohorts. Cohort 1 will consist of 32 healthy subjects, and Cohort 2 will consist of 52 healthy subjects. Subjects in each cohort will receive 2 doses of IPI under fasted conditions in a 2-period, 2-sequence crossover design. Dosing in Period 1 and Period 2 will be separated by at least 7 days.

Part 2 is a 2-period, 2-sequence crossover design to assess the effect of a high-fat meal on the PK of the IPI-145 in 20 subjects. Subjects will receive single oral doses under fed (high-fat meal) and fasted conditions, separated by at least 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of non-child bearing potential between 18-50 years of age
* Body Mass Index (BMI): 18.0 - 32.0 kg/m2.
* Healthy subjects: in good health, determined by no clinically significant findings from clinical evaluations
* Provided written informed consent prior to any study specific procedures

Exclusion Criteria:

* Women of childbearing potential
* Healthy subjects: positive screening test for hepatitis B surface antigen, hepatitis C antibody, or HIV-1/HIV-2 antibodies
* ECG at screening showing QTcF ≥ 450 msec
* Evidence of clinically significant medical conditions
* History of gastrointestinal disease or surgery that may affect drug absorption
* Positive T-Spot (tuberculosis)TB test at screening
* Any active infection at the time of screening or admission

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Assessment of bioequivalence of the IPI-145 test and reference formulations | 24 Hours
Pharmacokinetic Parameter (AUClast ) of IPI-145 | Over 24 hours
Pharmacokinetic Parameter (AUCinf ) of IPI-145 | Over 24 hours
Pharmacokinetic Parameter (Cmax) of IPI-145 | Over 24 hours

SECONDARY OUTCOMES:
Incidence of adverse events following administration of IPI-145 | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (1):
- Lenexa, Kansas, United States